CLINICAL TRIAL: NCT06867029
Title: Comparative Study Between Onlay and Sublay Mesh in Treatment of Ventral Hernia
Brief Title: Onlay and Sublay Mesh in Treatment of Ventral Hernia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mohamed Beloul Ali, Resident of General Surgery, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mohamed Beloul
Record Dates: First submitted 2025-03-05; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2023-05

CONDITIONS: Ventral Hernia
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Active Comparator): About 15 patients subjected to ventral hernia of onlay mesh procedure (mesh on external oblique muscle)
  Interventions: Procedure: Onlay Mesh
- Group II (Active Comparator): About 15 patients subjected to ventral hernia of sublay mesh procedure (mesh in the retromuscular space)
  Interventions: Procedure: Onlay Mesh

INTERVENTIONS:
Procedure: Onlay Mesh — to compare between two techniques of mesh placement in uncomplicated ventral hernias, onlay (mesh on external oblique) versus sublay (mesh in the retromuscular space).
  Other Names: Sublay Mesh

SUMMARY:
Hernia is defined as aprotrusion of viscus or part of viscus usually within a peritonial sac through a defect in the abdominal wall.

Ventral abdomenal hernias include all the hernias occuring through the anterior abdominal wall excluding groin hernias ( incisinal hernia, epigastric hernias, paraumbilical hernias, umbilical and lumbar hernias)

DETAILED DESCRIPTION:
Ventral hernia can be categorized according to their characteristic into reducible, irreducible or incarcerated , strangulated and recurrant ventral hernia.

The cause of a primary ventral hernia ia s far from completely understood, but it is undoubtedly multifactorial. familial prediposing play a role with increasing evidance of connective tissue disorders, they are considered as a leading cause of abdominal surgery and account for 2-10% of all abdomenal wall hernias .

Clinical data show that 52% of incisional hernias occur within 6 months postoperative as a result of excessive tension and inadeqate healing of aprevious incision.

The history of prothetic repair in abdominal wall hernias began in 1844 within the use of silver wire coils placed in the floor of groin to induce an inflammatory fibrosis . meny prosthetic material have been tried in hernia repair, but the two most common in current use are polypropylene mesh and expanded polytetrafluoroethylene.

The repair of ventral hernia varies from primary closure, primary closure with an onlay mesh reinforcement, sublay mesh placement, and intraperitonial mesh placement. Primary closure techniques are usually performed for smal fascial defects less than 5 cm in the greaters diameter

An onlay , usually of polyproptlene mesh is sutured to the anterior rectus sheeth after the fascial defect has been closed primary, thes type of repair has the potential advantage of keeping the mesh separeted from the abdomenal content by full abdominal muscle fascial wall thikness.

The sublay (retrorectus) placement of mesh, became popular in 1990, the recurence rates with this repair have been stated to be less than 10%.

ELIGIBILITY:
Inclusion Criteria:

* Ventral Hernia patients

Exclusion Criteria:

* Age below 18 years.
* Complicated hernia.
* Uncompensated heart or lung diseases, haemorrhagic disorders

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-05-10 (Actual); Primary Completion 2024-07-05 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
Post operative Pain | 4 hours post operative
  Assessment of post operative Pain by VAS scale

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Hassan, Professor, Study Chair — General Surgery, Faculty of Medicine, Al Azhar University, Assiut
Locations (1):
- Al-Azhar University Hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided